CLINICAL TRIAL: NCT02005029
Title: Erythromycin in Parkinson's Disease: A Pilot Study of Its Effects on Levodopa Pharmacokinetics and Pharmacodynamics
Brief Title: Erythromycin in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HM15105
Record Dates: First submitted 2013-09-18; First posted 2013-12-09 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson's Disease; Levodopa
Keywords: Parkinson's Disease; Levodopa; motor fluctuations; gastroparesis
MeSH Terms: conditions — Parkinson Disease; Gastroparesis | interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): One time IV dose of placebo
  Interventions: Drug: placebo
- Erythromycin (Experimental): One time IV dose of 100 mg Erythromycin
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin
  Arms: Erythromycin
Drug: placebo
  Arms: Placebo

SUMMARY:
Gastroparesis (slow stomach emptying) is a common feature of Parkinson's Disease. Levodopa (Sinemet), a common medication for Parkinson's Disease, can make gastroparesis worse. Gastroparesis effects how the levodopa is absorbed and used by the body. This study will explore the possibility of using Erythromycin, a drug commonly used (off label) for gastroparesis, along with levodopa to determine if there is improved levodopa absorption and motor function.

DETAILED DESCRIPTION:
Participants will be required to make four visits for evaluation. Visit 1 is a screening visit, participants will receive the study drug or a placebo during visits 2 and 3, and visit 4 is a follow up visit. Participants will provide blood and urine samples during the visits. Participants will also be required to complete questionnaires and a series of motor tests.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a definitive diagnosis of Parkinson's Disease (per United Kingdom brain bank criteria), Hoehn and Yahr stage 1-3,
* must exhibit unequivocal levodopa responsiveness
* must be able to distinguish between the "off" versus "on" state
* Subjects must be on a stable dose of levodopa for at least 28 days prior to enrollment and should be anticipated to maintain a stable dose throughout both study periods
* Subjects may be on concomitant therapy with Monoamine oxidase B inhibitors, entacapone, and amantadine, though the doses of these medications must have remained stable for at least 28 days prior to enrollment and must be expected to remain stable throughout both study periods.

Exclusion Criteria:

* History of deep brain stimulation for Parkinson Disease
* History of ablative (tissue removal) surgery for Parkinson Disease
* Presence of dementia (MMSE<25)
* Presence of active psychosis
* History of any chronic gastrointestinal diseases
* History of any prior gastrointestinal surgeries except for appendectomy, cholecystectomy, and hysterectomy
* Any gastrointestinal surgeries in the past 3 months
* Severe dysphagia (difficulty swallowing) to pills or food
* History of physiological or mechanical gastrointestinal obstruction
* History of strictures or fistulae (abnormal or narrow connections) along the gastrointestinal tract
* History of gastric bezoars (undigested mass)
* Allergy to wheat, soy, milk, or nuts
* Presence of portable electromechanical devices such as pacemaker, defibrillator, or infusion pump
* Female subjects who are pregnant or lactating
* Symptomatic orthostatic hypotension (low blood pressure)
* Diabetes
* Presence of symptomatic anemia
* Abnormal liver or kidney function
* Cardiac arrhythmia (past or present) or abnormal QT interval on entrance EKG
* Known hypersensitivity to any of the study drugs
* Subjects receiving certain medications during specified time frames

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Cloud, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Parkinson's Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen patients were screened for eligibility between April 2013 and June 2015 at the Virginia Commonwealth University Parkinson's and Movement Disorders Center.
Pre-assignment Details: 10 of 18 participants were randomized. Of those not randomized, 7 did not meet eligibility criteria and 1 was withdrawn by the principal investigator prior to randomization due to noncompliance with the protocol.
Groups:
- Placebo First Then Erythromycin: One time IV dose of placebo followed by 1 time IV dose of Erythromycin (after 2 week washout)
- Erythromycin Then Placebo: One time IV dose of 100 mg Erythromycin followed by 1 time IV dose of placebo (after 2 week washout)
Period: First Intervention (1 Day)
Arm/Group | Placebo First Then Erythromycin | Erythromycin Then Placebo
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — participant withdrawn for noncompliance | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Placebo First Then Erythromycin | Erythromycin Then Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo First Then Erythromycin | Erythromycin Then Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First Then Erythromycin | Erythromycin Then Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [51 to 77] | 64.0 [50 to 76] | 64.3 [50 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Time
Description: Mean gastric emptying time in minutes as measured by SmartPill
Time Frame: 2 weeks, between visits 2 and 3
Population: Of the original ten participants; one participant's data was excluded due to symptomatic orthostasis which likely confounded her results, one participant was withdrawn early due to noncompliance, and four participants were unable to complete a SmartPill evaluation.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Erythromycin: Mean gastric emptying time for participants receiving erythromycin
- Placebo: Mean gastric emptying time for participants receiving placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 4 | 4
minutes | 105 (66.5) | 180 (40.6)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.036, t-test, 2 sided

2. Primary Outcome: Area Under the Curve 0-4 Hours for Plasma Levodopa After Erythromycin Versus Placebo
Description: Mean Area under the Curve 0-4 hours for plasma levodopa after erythromycin versus placebo. Plasma samples were collected at the following times post-levodopa dose: 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, and 240 minutes.
Time Frame: 2 weeks, between visits 2 and 3
Population: Of the original ten participants; one participant's data was excluded due to symptomatic orthostasis which likely confounded her results, one participant was withdrawn early due to noncompliance, and one participant had undetectable plasma levodopa levels through out the study and was thus excluded from the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL*min
Groups:
- Erythromycin: Area under the curve 0-4 hours for plasma levodopa after erythromycin
- Placebo: Area under the curve 0-4 hours for plasma levodopa after placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 7 | 7
ng/mL*min | 123237 (137561) | 103584 (106271)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; Erythromycin:Placebo AUC ratio = 1.07, Standard Deviation 0.43

3. Secondary Outcome: 9-hole Peg Test Right Hand
Description: Change in motor function as assessed by 9-hole peg test for upper extremity manipulation/dexterity. This test measures the total time required to place and remove 9 holes in a pegboard. Each hand is tested separately.
Time Frame: 2 weeks, between visits 2 and 3
Population: Of the original 10 participants, one participant's data was excluded due to symptomatic orthostasis which likely confounded her results and one participant was withdrawn early due to noncompliance.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Erythromycin: Mean time for right hand after erythromycin
- Placebo: Mean time for right hand after placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 25.36 (4.37) | 25.80 (4.23)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

4. Secondary Outcome: 9-hole Peg Test Left Hand
Description: as for outcome 3
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 29.36 (6.27) | 27.33 (6.45)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

5. Secondary Outcome: Five Times Sit-to-stand Test
Description: Change in motor function as measured by Five times sit-to-stand test. This test measures the total time to complete 5 repetitions of sit to stand.
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Erythromycin: Five times sit-to-stand for all participants receiving erythromycin
- Placebo: Five times sit-to-stand for all participants receiving placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 11.09 (2.24) | 10.09 (2.48)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.4405, t-test, 2 sided

6. Secondary Outcome: Comfortable 20 Feet Gait Speed (CGS)
Description: Change in motor function as assessed by comfortable 20 feet gait speed (CGS)
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Erythromycin: Mean CGS for all participants receiving erythromycin
- Placebo: Mean CGS for all participants receiving placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 4.26 (0.44) | 4.10 (0.69)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.6011, t-test, 2 sided

7. Secondary Outcome: Timed up and go Test (TUAG) Comfortable Speed
Description: Change in motor function as assessed by timed up and go test (comfortable speed). This test measures the total time to stand from a chair, walk 10 feet, and return to sitting.
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Erythromycin: TUAG (comfortable speed) after erythromycin
- Placebo: TUAG (comfortable speed) after placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 8.67 (1.33) | 8.26 (1.05)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.8923, t-test, 2 sided

8. Secondary Outcome: Timed up and go Test (TUAG) Fast Speed
Description: Change in motor function as assessed by timed up and go test (fast speed). This test measures the total time to stand from a chair, walk 10 feet, and return to sitting.
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Erythromycin: TUAG (fast speed) after erythromycin
- Placebo: TUAG (fast speed) after placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
seconds | 6.79 (0.927) | 6.85 (1.06)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.832, t-test, 2 sided

9. Secondary Outcome: Change in Dyskinesia
Description: Mean total AIMS (Abnormal Involuntary Movements Scale) score after receiving erythromycin minus mean total AIMS score after receiving placebo. The AIMS test has a total of twelve items rating involuntary movements of various areas of the patient's body. Ten of the items are rated on a five-point scale of severity from 0-4. The scale is rated from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe). Two of the items are not scored. Total score range is from 0 to 40. Higher scores represent more severe dyskinesia (a worse outcome).
Time Frame: 2 weeks, between visits 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Erythromycin: AIMS after receiving erythromycin
- Placebo: AIMS after receiving placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
units on a scale | 0.875 (1.458) | 0.375 (1.061)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.1546, t-test, 2 sided

10. Secondary Outcome: MDS-UPDRS Part 3 (Movement Disorders Society- Unified Parkinson's Disease Rating Scale)
Description: Part 3 of this scale is a standardized physical assessment that quantifies the total burden of motor symptoms in Parkinson's disease patients. Each of the 18 items on the scale is rated from 0 (none, 1 (slight), 2 (mild), 3 (moderate) and 4 (severe). Scores range from 0-72. Higher scores represent a more severe burden of motor symptoms (a worse outcome).
Time Frame: 2 weeks, between visits 2 and 3
Population: One participant's data was excluded due to symptomatic orthostasis which likely confounded her results and one participant was withdrawn early due to noncompliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 8 | 8
units on a scale
  Before or "off" levodopa | 30.75 (13.26) | 25.37 (11.09)
  After or "on" levodopa | 17.13 (11.48) | 16.50 (8.38)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.0314, t-test, 2 sided; Mean Difference (Final Values) = 4.75, Standard Deviation 5.00 — Mean difference in "on" score versus "off" score from the MDS UPDRS Part 3 on day of erythromycin minus the mean difference in 'on" score versus "off" score on day of placebo

11. Secondary Outcome: Mean Cmax of Plasma Levodopa After Erythromycin Versus Placebo
Description: Mean Cmax of plasma levodopa after erythromycin versus placebo. Plasma samples were collected at the following times post-levodopa dose: 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, and 240 minutes.
Time Frame: 2 weeks, between visits 2 and 3
Population: Of the original ten participants; one participant's data was excluded due to symptomatic orthostasis which likely confounded her results, one participant was withdrawn early due to noncompliance, and one participant had undetectable plasma levodopa levels throughout the study and was thus excluded from the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Erythromycin: Cmax of plasma levodopa after erythromycin
- Placebo: Cmax of plasma levodopa after placebo
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 7 | 7
ng/mL | 1267 (1012) | 1395 (1015)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; Erythromycin:Placebo Cmax ratio = 0.83, Standard Deviation 0.24

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Description: Participants were followed from the beginning to the end of their active participation or the resolution of any adverse events.
Groups:
- Erythromycin: Participants who received a one time dose of IV erythromycin
- Placebo: Participants who received a one time dose of placebo
Arm/Group | Erythromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 4/9 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythromycin (N=9) | Placebo (N=10)
symptomatic orthostasis (Cardiac disorders) | 1 (1) | 1 (1) — One participant developed symptomatic orthostatic hypotension during both her erythromycin and placebo dosing days. This resolved within a few minutes following sips of water and rest.
akathisia (Nervous system disorders) | 1 (1) | 0 (0) — One participant developed self limited akathisia after taking levodopa during his erythromycin dosing day. This resolved after a few minutes with no intervention.
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — One participant developed a single episode of loose stool during her erythromycin dosing day. No intervention was necessary.
possible hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) — One participant had trace hematuria on urinalysis from his final safety visit (occurring after his erythromycin dosing day). Urinalysis was repeated by primary care provider one day later and was normal.
transaminitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — One participant had a mild transaminitis identified at his final safety visit (after placebo dosing day). This was thought to be due to over use of pain medication for an acute back injury. This resolved after stopping pain medication.

LIMITATIONS AND CAVEATS:
An overall limitation was the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes